CLINICAL TRIAL: NCT03263871
Title: Pilot Study of PTM202 for the Treatment of Environmental Enteric Dysfunction (EED)
Brief Title: PTM202 for the Treatment of Environmental Enteric Dysfunction (EED)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19993
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Environmental Enteric Dysfunction
Keywords: nutrition

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): PTM202 and micro-nutrient sprinkles
  Interventions: Dietary Supplement: PTM202; Dietary Supplement: micro-nutrient sprinkles
- Control (Other): micro-nutrient sprinkles
  Interventions: Dietary Supplement: micro-nutrient sprinkles

INTERVENTIONS:
Dietary Supplement: PTM202 — PTM202 given twice daily for 30 days.
  Arms: Intervention
Dietary Supplement: micro-nutrient sprinkles — Micro-nutrient sprinkles will be given twice daily for 30 days.

SUMMARY:
The purpose of this study is to assess the effectiveness of PTM202 in treating environmental enteric dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 - 9 months old
* -1> Weight-for-age Z score > -3
* Parental consent to participate and receive daily supplementation with either PTM202 and/or micro-nutrient sprinkles, participate in specimen collection

Exclusion Criteria:

* Presence of known kidney, liver, heart, developmental, or neurologic disease
* Allergy to milk and/or egg (assessed by history)
* Milk intolerance (assessed by history)
* Abnormal liver or kidney function tests
* Family is planning to move from the study area or children is enrolled to the other clinical trial within 3 months of follow up
* Child being exclusively breast fed at the time of enrollment

Ages: 6 Months to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2017-10-14 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
EED biomarker composite score | 4 months
  composite score of fecal Reg 1B, fecal myeloperoxidase, urinary lactulose: mannitol ratio, serum soluable-CD14, and serum C-reactive protein

SECONDARY OUTCOMES:
Weight gain | 4 months
Height gain | 4 months
Number of diarrheal episodes | 4 months
Glucose hydrogen breath test | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No